CLINICAL TRIAL: NCT04453124
Title: An Accessible Low-cost Plant Treatment for Cutaneous Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oriol Mitja (Other)
Collaborators: The University of Papua New Guinea (Unknown); The Royal Botanic Gardens, Kew (Unknown)
Responsible Party: Sponsor-Investigator, Oriol Mitja, Dr. Oriol Mitja, Lihir Medical Centre
Organization: Lihir Medical Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAPKOKOPO
Record Dates: First submitted 2020-06-21; First posted 2020-07-01 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Yaws; Cutaneous; Cutaneous Ulcer; Yaws
MeSH Terms: conditions — Yaws; Skin Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor of healing outcomes through pictures will not know the arm of origen of the pictures .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Soap and Water (No Intervention): Standard of care using soap and water
- Ficus Septica Sap (Experimental): Ficus Septica Sap, topical cream, 50ul, daily, for 2 days
  Interventions: Biological: Topical antiseptic treatment
- Chlorhexidine (Topical) (Active Comparator): Chlorhexidine, topical solution, 50ul, daily, for 2 days
  Interventions: Biological: Topical antiseptic treatment

INTERVENTIONS:
Biological: Topical antiseptic treatment — Prevent the development of bacterial cutaneous ulcers by applying antiseptic sap from Ficus septica tree on small wounds.
  Arms: Chlorhexidine (Topical); Ficus Septica Sap

SUMMARY:
In a search for accessible treatment options, plant medicines used by different communities in Papua New Guinea have been tested to identify the sap of the tree, Ficus septica, as a promising antibacterial agent in vitro.

This is an open label clinical trial using an interventional approach, to compare the effect of the antiseptic plant sap and standard topical antiseptic, on the rate of wound development prevention and bacterial growth. If shown to be effective, this readily available plant medicine can provide a zero-cost treatment option in remote areas of PNG.

DETAILED DESCRIPTION:
The cutaneous ulcer is a painful and debilitating bacterial infection that is common in rural areas of Papua New Guinea (PNG). Systematic treatment with topical antiseptics such as chlorhexidine cream in theory represents a viable treatment option, but in reality, effective treatment of cutaneous ulcers in Papua New Guinea is greatly hindered by the remote and highly inaccessible areas that affected communities often live in. In a search for more accessible treatment options, plant medicines used by different communities in Papua New Guinea have been tested to identified the sap of the tree, Ficus septica, as a promising antibacterial agent in vitro. The sap displays comparable activity to chlorhexidine in disc diffusion assays with gram-positive bacterial wound pathogens. It also appears to dampen the pro-inflammatory responses of neutrophils by down regulating interleukin-6 expression. The sap forms a flexible plastic-like wound covering which may help deter flies from feeding on the wounds, and unlike chlorhexidine cream, the Ficus tree is easy to find where affected communities live. For this reason, this study aims to perform an open label clinical trial using an interventional approach, to compare the effect of this antiseptic plant sap and of a standard topical antiseptic, on the rate of wound development prevention and bacterial growth. If shown to be effective, this readily available plant medicine can provide a zero-cost treatment option in remote areas of PNG.

ELIGIBILITY:
Inclusion Criteria:

-children aged 5 to 15 with parental consent and with one or more skin breaks of any nature (i.e. Skin cuts, scratch, scrapes or abrasion and mosquito bites) that are less than 1cm in major diameter. Written informed consent by parent or guardian will be required before enrolment.

Exclusion Criteria::

* All participants who have received medical treatment for skin ulcers up to 2 months prior to recruitment (azithromycin, amoxicillin, benzathine penicillin, etc.).
* Patients who require antibiotic treatment for another condition not-related to the study.
* Known history of hypersensitivity, allergic or adverse reaction to the study product.
* Patients presenting cutaneous ulcer more than 1cm

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with Clinical Healing in each arm | 21 days
  surface reduction by more than 50%
Number of participants with Clinical Healing in each arm | 21 days
  Ulcer healing determined by a professional dermatologist, described as as: appearance of granulation tissue, healed borders, dry ulcer, no exudation.

SECONDARY OUTCOMES:
Changes in wound microbiology | 21 days
  Up to five key pathogens identified by next generation sequencing of wound fluids will be quantified at Day 0 and at Day 21 for samples from each arm of the study

CONTACTS AND LOCATIONS:
Locations (2):
- Papua New Guinea (2):
  - Lihir Medical Centre, Londolovit, New Ireland Province
  - University of Papua New Guinea, Port Moresby

IPD SHARING:
Plan to Share IPD: Yes
All individual variables will be available through direct contact with corresponding author
Supporting Information: Study Protocol
Time Frame: After publication of data for 1 year